CLINICAL TRIAL: NCT05887882
Title: A Phase I Study of Intra-Tumoral Injections of Ex Vivo Expanded Natural Killer Cells in Children and Young Adults With Recurrent or Progressive Malignant Brain Tumors
Brief Title: Intra-Tumoral Injections of Natural Killer Cells for Recurrent Malignant Pediatric Brain Tumors
Acronym: PNOC028
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sabine Mueller, MD, PhD (Other)
Collaborators: Rally Foundation (Unknown); Washington University School of Medicine (Other); Nationwide Children's Hospital (Other); CureSearch (Unknown); Tommy Strong Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Sabine Mueller, MD, PhD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 210831; NCI-2023-03216 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Brain Tumor; Recurrent Pediatric Brain Tumor; Pediatric Neoplasm
Keywords: Transforming growth factor beta imprinted; Natural Killer Cells
MeSH Terms: conditions — Neoplasms | interventions — Cell Count; Drug Implants; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level 2 (3x10^6) - Starting Dose (Experimental): Enrolled participants must proceed to surgery for tumor resection and Ommaya placement into the resection cavity within 14 days of enrollment. Starting dose of 3x10^6 of TGFβi NK cells (first dose) may be administered at least 14 days after the Ommaya reservoir placement and may not start until all acute surgical complications have resolved (maximum of 6 weeks after enrollment). TGFβi NK cell infusions through the Ommaya reservoir will occur once weekly for three weeks followed by one rest week. If participants have stable or improved disease, participants may continue to receive therapy for a total of 3 cycles.
  Interventions: Biological: Universal Donor (UD) Transforming growth factor beta imprinting (TGFβi) Natural Killer (NK) Cells; Procedure: Implantation; Procedure: Magnetic Resonance Imaging (MRI); Other: Quality-of-Life Assessment
- Dose Level 3 (3x10^7) (Experimental): If no safety or toxicity events are demonstrated by the starting dose cohort, enrolled participants in the next dosing cohort must proceed to surgery for tumor resection and Ommaya placement into the resection cavity within 14 days of enrollment. The dose of 3x10^7 of TGFβi NK cells (first dose) may be administered at least 14 days after the Ommaya reservoir placement and may not start until all acute surgical complications have resolved (maximum of 6 weeks after enrollment). TGFβi NK cell infusions through the Ommaya reservoir will occur once weekly for three weeks followed by one rest week. If participants have stable or improved disease, participants may continue to receive therapy for a total of 3 cycles.
  Interventions: Biological: Universal Donor (UD) Transforming growth factor beta imprinting (TGFβi) Natural Killer (NK) Cells; Procedure: Implantation; Procedure: Magnetic Resonance Imaging (MRI); Other: Quality-of-Life Assessment
- Dose Level 4 (3x10^8) (Experimental): If no safety or toxicity events are demonstrated by the previous dose cohort, enrolled participants in the next dosing cohort must proceed to surgery for tumor resection and Ommaya placement into the resection cavity within 14 days of enrollment. The dose of 3x10^8 of TGFβi NK cells (first dose) may be administered at least 14 days after the Ommaya reservoir placement and may not start until all acute surgical complications have resolved (maximum of 6 weeks after enrollment). TGFβi NK cell infusions through the Ommaya reservoir will occur once weekly for three weeks followed by one rest week. If participants have stable or improved disease, participants may continue to receive therapy for a total of 3 cycles.
  Interventions: Biological: Universal Donor (UD) Transforming growth factor beta imprinting (TGFβi) Natural Killer (NK) Cells; Procedure: Implantation; Procedure: Magnetic Resonance Imaging (MRI); Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Universal Donor (UD) Transforming growth factor beta imprinting (TGFβi) Natural Killer (NK) Cells — The TGFβi NK cell product will be manufactured in the Cell Therapy Laboratory at Nationwide Children's Hospital and given via infusion.
  Other Names: UD TGFβi NK cells; UD TGFβi NK cell product
Procedure: Implantation — Undergo placement of Ommaya reservoir
Procedure: Magnetic Resonance Imaging (MRI) — Imaging procedure
  Other Names: MRI
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: QOL Assessment

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of ex vivo expanded natural killer cells in treating patients with cancerous (malignant) tumors affecting the upper part of the brain (supratentorial) that have come back (recurrent) or that are growing, spreading, or getting worse (progressive). Natural killer (NK) cells are immune cells that recognize and get rid of abnormal cells in the body, including tumor cells and cells infected by viruses. NK cells have been shown to kill different types of cancer, including brain tumors in laboratory settings. Giving NK cells from unrelated donors who are screened for optimal cell qualities and determined to be safe and healthy may be effective in treating supratentorial malignant brain tumors in children and young adults.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of natural killer (NK) cells that have been propagated ex vivo with genetically-modified feeder cells and administered intra-tumoral via an Ommaya reservoir in participants with recurrent or progressive malignant brain tumors.

II. To determine the recommended phase 2 dose (RP2D) for natural killer (NK) cells that have been propagated ex vivo with genetically-modified feeder cells and administered intra-tumoral via an Ommaya reservoir in participants with recurrent or progressive malignant brain tumors.

EXPLORATORY OBJECTIVES:

I. To determine the 6 months overall survival (OS), defined as the percentage of participants in the study who are alive at 6 months following start of treatment.

II. To determine the persistence, immuno-phenotype and function of adoptively-transferred expanded NK cells and correlate the findings with the overall response.

III. To determine the immune signature-based profile of each patient's tumor. IV. To determine changes in the T-cell receptor (TCR) repertoire diversity before and after Transforming growth factor beta imprinted (TGFβi) NK cell treatment.

V. To evaluate the effect of systemic steroids on the persistence and efficacy of TGFβi NK cells.

VI. To assess Quality of Life (QOL) and cognitive measures in children and young adults with recurrent or progressive malignant brain tumors.

VII. To assess patient and/or proxy satisfaction with study participation via patient-reported outcome (PRO) measures in the context of race ethnicity and other health related social risks.

VIII. To assess on therapy toxicity in the context of race, ethnicity and other health related social risks.

OUTLINE: This is a dose-escalation study.

Participants undergo placement of an Ommaya reservoir and receive universal donor expanded TGF-beta-imprinted NK cells (TGFBi NK cells) intratumorally over 5 minutes via Ommaya reservoir on day 1 of each cycle. Cycles repeat every 28 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Participants also undergo magnetic resonance imaging (MRI) of the brain during screening and on study and collection of tumor-associated fluid via Ommaya reservoir on study. Participants may also undergo MRI of the spine and lumbar puncture as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a histologically-confirmed recurrent or progressive malignant brain tumor including, but not limited to, infant-type hemispheric glioma, gliosarcoma, intracranial sarcoma and WHO Grade II ependymoma.
2. Participants should be candidates for resection of the recurrent tumor and be deemed candidate for placement of an Ommaya reservoir placed intra-cavitary/intra-tumoral; measurable residual tumor after surgery is not required for study entry. Pre-operative imaging needs to estimate that the resection cavity will be at least 2 cm x 2 cm in two dimensions for participants to be eligible.
3. Given the lack of a standard of care treatment for children with recurrent or progressive malignant brain tumors, participants must have completed first-line treatment with radiation and/or chemotherapy prior to participating in this trial if applicable.
4. All participants must be ≥ 1 year of age and ≤ 39 years of age at the time of entry into the study. The first 3 participants must be ≥ 8 years of age and ≤ 39 years of age at the time of entry into the study.
5. Performance Score: Karnofsky ≥ 50 for participants > 16 years of age and Lansky ≥ 50 for participants ≤ 16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
6. Must have recovered from the acute toxic effects of prior therapy (i.e., NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5, grade 1 or less)

   * An interval of at least 12 weeks must have elapsed since the completion of radiation therapy.
   * Chemotherapy/biologic therapy: All cytotoxic chemotherapy/biologic therapy must be discontinued ≥ 7 days prior to enrollment (except 3 weeks for temozolomide and 6 weeks from last dose of nitrosoureas)
   * Immunotherapy: The last dose of anti-tumor antibody therapy must be at least 3 half-lives or 30 days, whichever is shorter, from the time of enrollment
   * For targeted agents only, participants should have recovered from any toxicity of the agent and have a minimum of 2 weeks since the last dose.
   * For participants who have received prior bevacizumab, at least 4 weeks is required.
7. Organ Function Requirements:

   1. Adequate Bone Marrow Function Defined as:

      * Peripheral absolute neutrophil count (ANC) >750/mm^3.
      * Platelet count >75,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to registration).
   2. Adequate Renal Function Defined as:

      * A serum creatinine ≤ 1.5 x upper limit normal (ULN) based on age/gender.
   3. Adequate Liver Function Defined as:

      * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age; in presence of Gilbert's syndrome, total bilirubin ≤ 3 x ULN or direct bilirubin ≤ 1.5 x ULN.
      * Alanine aminotransferase (ALT) ≤ 3 x ULN.
      * Aspartate aminotransferase (AST) ≤ 3 x ULN.
   4. Adequate Neurologic Function Defined as:

      * Participants with seizure disorder may be enrolled if seizures are well-controlled. Participants on non-enzyme inducing anticonvulsants may be excluded pending interaction(s) with study drug.
      * Signs and symptoms of neurologic deficit must be stable for ≥ 1 week prior to registration.
8. The effects of Transforming growth factor beta resistant (TGFβi) natural killer (NK) cells on the developing human fetus are unknown. For this reason and because TGFβi NK cells as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 6 months after completion of TGFβi NK cells administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
9. Participants must enroll on PNOC COMP if PNOC COMP is open to accrual at the enrolling institution
10. A legal parent/guardian or patient must be able to understand, and willing to sign, a written informed consent and assent document, as appropriate.
11. Corticosteroids: Participants who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration. The patient steroid dose should be no more than a steroid-equivalent of dexamethasone 0.1 mg/kg/day (or maximum 4 mg/day; whichever is the lower dose) at time of enrollment.

Exclusion Criteria:

1. Tumor involvement that would require ventricular or brainstem injection or access through a ventricle or significant risk of ventricular penetration in order to deliver the TGFβi NK cells.
2. Participants undergoing needle or open biopsy.
3. Participants who are receiving any other investigational agents.
4. Women of childbearing potential must not be pregnant or breast-feeding.
5. Evidence of active uncontrolled infection or unstable or severe intercurrent medical conditions.
6. Any medical condition that precludes surgery.
7. Prothrombin time/international normalized ratio (PT/INR) or partial thromboplastin time (PTT) > 1.5 x ULN.
8. Participants with a known disorder that affects their immune system, such as human immunodeficiency virus (HIV), or an auto- immune disorder requiring systemic cytotoxic or immunosuppressive therapy are not eligible.
9. Evidence of bleeding diathesis or use of anticoagulant medication or any medication which may increase the risk of bleeding. If the medication can be discontinued >1 week prior to NK cell infusion then the subject may be eligible following consultation with the Study Chairs.
10. Participants with significant systemic or major illnesses including but not limited to: congestive heart failure, ischemic heart disease, kidney disease or renal failure, organ transplantation, or significant psychiatric disorder.
11. History or current diagnosis of any medical or psychological condition that in the Investigator's opinion, might interfere with the participants ability to participate or inability to obtain informed consent because of psychiatric or complicating medical problems.

Important note: The eligibility criteria listed above are interpreted literally and cannot be waived.

Ages: 1 Year to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment-emergent adverse events | From initiation of study treatment until 30 days from the end of therapy, approximately 1 year
  Adverse events and clinically significant laboratory abnormalities (meeting grade 3, 4, or 5 criteria according to NCI CTCAE) will be summarized by maximum intensity and relationship to study drug(s). Grade 1 and 2 adverse events will be summarized if related to study therapy. Descriptive statistics will be utilized to display the data on toxicity seen. Toxicities will be summarized by tabulation in terms of type, grade and attribution for each dose level of each group of patients studied at the end of the trial.
Recommended Phase II dose (RP2D) | From initiation of study treatment until 30 days from the end of therapy, approximately 1 year
  RP2D is defined as the dose level at which fewer than one-third of participants experience a dose limiting toxicity (DLT)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (6):
- United States (6):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins, Baltimore, Maryland
  - Washington University in Saint Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data may be shared with collaborating researchers.
Supporting Information: Study Protocol